CLINICAL TRIAL: NCT05394545
Title: A Randomized, Phase II, Open-Label Study Evaluating the Nu-V3 Cranial Nerve Stimulation Treatment Device in Patients With Chronic Pain, Anxiety, Depression, and/or Sleeplessness
Brief Title: Phase II Trial of Nu-V3 Non-Invasive Nerve Stimulation Device for Chronic Pain, Anxiety, Depression, Sleeplessness
Acronym: Nu-V3P2RCT
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: staffing challenges
Sponsor: Nu-Life Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Nu-V3 RCT Protocol
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Chronic Pain; Anxiety; Depression; Sleeplessness
Keywords: Device; TENS; Neuromodulation; PTSD; Neuropathy; Inflammatory; Arthritis; Chronic Pain; Fibromyalgia; Osteoarthritis; TMJ; Insomnia
MeSH Terms: conditions — Chronic Pain; Anxiety Disorders; Depression; Sleep Initiation and Maintenance Disorders; Stress Disorders, Post-Traumatic; Arthritis; Fibromyalgia; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: A Randomized, Phase II, Open-Label Study Evaluating the Nu-V3 Cranial Nerve Stimulation Treatment Device in Patients with Chronic Pain, Anxiety, Depression, and/or Sleeplessness
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Nu-V3 treatment arm (Experimental): Treatment with the Nu-V3 Device.
  Interventions: Device: Nu-V3
- Observation treatment arm (SOC, control) (No Intervention): Observation following stable standard of care.

INTERVENTIONS:
Device: Nu-V3 — The Nu-V3 device provides a continuous flow of intermittent, low frequency electrical pulses to the ear's specific cranial nerve endings. This treatment is delivered 24 hours a day for the first 12 weeks, then is delivered two weeks on, one week off for the following 12 weeks.
  Arms: Nu-V3 treatment arm

SUMMARY:
This Nu-V3 clinical study is a randomized, phase II, open-label study evaluating the Nu-V3 cranial nerve stimulation treatment device in patients with chronic pain, anxiety, depression, and/or sleeplessness.

DETAILED DESCRIPTION:
Subjects randomized to receive the Nu-V3 treatment will undergo the following regimen:

* At the baseline visit, patients will be asked to complete study questionnaires regarding all of the following symptoms: chronic pain, anxiety, depression, and/or sleeplessness, as well as their quality of life, active medications, medical history, and demographical information. The subject's primary symptom of concern will also be notated at baseline, for later assessment of continuation after week 12.
* At each subsequent visit, patients will be asked to complete study questionnaires regarding all the following symptoms: chronic pain, anxiety, depression, and/or sleeplessness, as well as their activity level and quality of life.
* The sessions will begin with the Nu-V3 device being clipped on the ear and three small pads (non-invasive) adhered to the surface of the ear. Each Nu-V3 device lasts for up to 28 days with a change in the pads approximately 7 days into the treatment.
* Each session takes approximately 15-20 minutes. The placement of the device takes approximately 5 minutes, and the remaining time is spent verifying ePRO form completion, and evaluating the patient for all device effects.
* The Nu-V3 device is mobile and is worn externally on the left ear 24 hours a day during treatment, fitting comfortably behind the ear. An electrical signal is sent to the external ear through coated wire leads attached to the device and adhesive pads which attach to three sites on the ear.
* Participants should be able to perform their typical day-to-day activities while wearing the device. They may shower while wearing the Nu-V3 device, if they do not get the device wet and use the small disposable ear covers that are provided for them.
* In the event the Nu-V3 gel pads are inadvertently removed or the device comes off, the participant will contact the site coordinator. The participant is encouraged to adjust the device placement as needed for comfort.
* Patients should not change their existing forms of treatment or medications without discussion with the study investigator.

Subjects randomized to the observation control arm of the study will undergo the following regimen:

* At the baseline visit, patients will be asked to complete study questionnaires regarding all the following symptoms: chronic pain, anxiety, depression, and/or sleeplessness, as well as their quality of life, active medications, medical history, and demographical information. The subject's primary symptom of concern will also be notated at baseline.
* At each subsequent visit, patients will be asked to complete study questionnaires regarding all the following symptoms: chronic pain, anxiety, depression, and/or sleeplessness, as well as their activity level and quality of life.
* Patients should not change their existing forms of treatment or medications without discussion with the study investigator.
* At completion of 12 weeks of standard of care treatment post study enrollment, observation (control arm) subjects will be offered a crossover into the treatment arm of the study for an additional 24 weeks.

Sample size For this Phase II study, a total of 100-200 subjects will be randomized 1:1 to either the Nu-V3 treatment arm or to the observation treatment arm (SOC, control).

Recruitment Participants are enrolled into relevant symptom cohorts based on their chronic pain, anxiety, depression, and/or sleeplessness symptom presentation at baseline and treated with the Nu-V3 device for 24 weeks.

Analyses Interim analysis of reported data will be based on baseline symptom cohort and conducted at 6, 12, 18, and 24 weeks during this time. The participant will be evaluated after the initial 12-week treatment period to assess for further therapeutic need. Upon having three consecutive weeks of mean symptom reduction of ≥70% via patient reported numerical scales, the participant will continue as described in the study assessments table, but without device therapy. Then if the participant's primary symptom score increases at any time by ≥20%, they may again continue device therapy until week 24, as depicted in section 4.1.

Study subjects randomized to the observation arm will be offered the opportunity to cross-over to the Nu-V3 study treatment arm upon completion of the initial 12-week observation study period.

ELIGIBILITY:
Inclusion Criteria:

* Participant is at least 18 years of age
* Participant presents with one or more of the following symptoms: chronic pain, anxiety, depression, and/or sleeplessness
* Participants must score greater than or equal to a 5/10 for their primary symptom score on the Baseline Symptom Questionnaire
* Patient's chosen primary symptom must have an available accrual slot for the participant. If patient scores greater than or equal to a 5/10 for a second symptom, they can be selected to accrue to another symptom slot.
* Participant has signed the Informed Consent Form

Exclusion Criteria:

* Participants with a hearing aid
* Participants with a pacemaker
* Participants with irregular heart rate or a heart rate lower than 60 beats per minute (bradycardia)
* Have had a transplant within the last 2 years
* Have had a heart attack or cardiac bypass surgery within the last 12 months
* Patients with complaints of dizziness or lightheadedness within the last 3 months
* Women who are pregnant
* Participants with Diabetic Retinopathy
* Current ear infection
* SBP < 100 and/or DBP < 60
* History of uncontrolled bipolar disorder within the last 12 months
* History of uncontrolled seizures within the last 12 months
* History of aneurysms
* History of syncope within the last 12 months
* Participants that have had a TIA or stroke within the last 12 months
* Participants with health problems deemed at risk for the study by the Principal Investigator
* Participants with any changes to Pain/Anxiety/Depression/Sleeplessness medications within last 60 days (participants that do not meet this medication- change washout period may be delayed until 60-day period is met)
* Participants that are currently under adjudication process for disability support, VA or other

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall safety from unanticipated problems or risks | Week 24
  At screening/baseline, a medical history will be obtained to capture relevant underlying conditions. The screening/baseline examinations will include BP, and HR. Baseline signs and symptoms are those that are assessed within 14 days prior to week 1 treatment.
  Concomitant medications will be collected from within 14 days prior to enrollment through the study treatment period and maintenance period.
  The primary safety endpoint is the occurrence of reported unanticipated problems involving risk to subjects or others ("UPIRTSOs"). These UPIRTSOs are defined as those problems which alter the risks to subjects or others. This includes any study suspensions or holds. The primary safety endpoint analyses will be based on a risk-benefit conclusion.
Effectiveness and overall change in reported primary symptom of concern: Chronic Pain | 12 and 24 weeks
  Chronic Pain - (PEG Scale) The PEG is a three-item instrument that measures pain intensity (one item) and pain interference (two items). The PEG is a three-item instrument that measures pain intensity (one item) and pain interference (two items). Each item is valued from 0 (no pain/interference) to 10 (as bad as you can imagine). The instrument score is calculated as the average of the three item values.
Effectiveness and overall change in reported primary symptom of concern: Anxiety | 12 and 24 weeks
  Anxiety - (GAD-7)The GAD-7 is a seven-item instrument that measures respondents' symptoms of anxiety. The GAD-7 is a seven-item instrument that measures respondents' symptoms of anxiety. Each item is scored on a four-point Likert scale, and values range from 0 ("Not at all") to 3 ("Nearly every day".) Items are summed to determine the instrument's score. Values of 10 or higher have been associated with moderate anxiety, while values of 15 or higher have been associated with severe anxiety.
Effectiveness and overall change in reported primary symptom of concern: Depression | 12 and 24 weeks
  Depression - (PHQ-9) The PHQ-9 is a nine-item instrument that measures depression-related symptoms and functional impairment. The PHQ-9 is a nine-item instrument that measures depression-related symptoms and functional impairment. Each item is scored on a four-point Likert scale and values range from 0 ("Not bothered at all") to 3 ("Bothered nearly every day.") The items' values are summed to determine the instrument's score. PHQ-9 values of 10 and 15 represent moderate and moderately severe depression respectively.
Effectiveness and overall change in reported primary symptom of concern: Sleeplessness | 12 and 24 weeks
  Sleeplessness - PROMIS short form 4a- This eight item instrument measures sleep disturbance and sleep-related impairment. This eight item instrument measures sleep disturbance and sleep-related impairment.

SECONDARY OUTCOMES:
Effectiveness: Symptom Frequency | 12 and 24 weeks
  In the Nu-V3 device treatment arm, the study will report the mean time from treatment initiation to reduction of symptoms of at least 30% in any of the four domains of symptom measurement.
Effectiveness: Symptom Severity | 12 and 24 weeks
  In both the Nu-V3 device treatment arm and the observation arm, the study will report the mean percentage change in symptoms severity from initiation to 12 and 24 weeks for each instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Vipul Kella, MD, Principal Investigator — Nu-Life Solutions
Locations (2):
- United States (2):
  - Greater Chicago Specialty Physicians (GCSP) - Schamuburg, Schaumburg, Illinois
  - EZ Clinic, Greenwood, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Nu-Life Solutions Homepage — https://www.nu-v3.com/

DOCUMENTS (2):
  • Study Protocol (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/45/NCT05394545/Prot_000.pdf
  • Informed Consent Form (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/45/NCT05394545/ICF_001.pdf